CLINICAL TRIAL: NCT04845932
Title: Finding Correlations Between Asthma Exacerbation, Physiological Measurements and Environmental Factors
Acronym: SCH Asthma
Status: Recruiting | Type: Observational
Sponsor: North Carolina State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Edgar Lobaton, Associate Professor - Dept. of Electrical and Computer Engineering, North Carolina State University
Other Study IDs: 16598
Record Dates: First submitted 2021-03-31; First posted 2021-04-15 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify asthma-related physiological changes observed by wearable devices in real-world conditions by monitor multiple sensing modalities (e.g., heart rate (HR), heart rate variability (HRV), activity level, spirometry, coughing sounds) in order to find reliable signatures of impending asthma exacerbation and systematically explore any challenges on the use of wearable technologies.

DETAILED DESCRIPTION:
The study aims to identify asthma-related physiological changes observed by wearable devices in real-world conditions. The investigators aim to monitor multiple sensing modalities (e.g., heart rate (HR), heart rate variability (HRV), activity level, spirometry, coughing sounds) in order to find reliable signatures of impending asthma exacerbation and systematically explore any challenges on the use of wearable technologies. A variety of off-the-shelf devices as well as the prototype HET platform developed by the NCSU ASSIST center will be used for data collection.

The investigators plan to engage adolescents (ages 14-18) for a period of up to four months of monitoring. They will be asked to wear the wrist monitoring device for at least 8 hours daily and chest monitoring devices for at least 12 hours a week, to take daily measurements using a spirometer, and answer weekly questionnaires online and virtual interviews (at 1-week,1-month and 3-months) about their asthma control and experiences with the devices.

Wearable devices are increasingly popular with young people and are capable of providing dynamically calculated up-to-the-minute measurements of a number of physiologic parameters, including heart rate, heart rate variability, respiratory rate, activity levels, and cough. The cough sounds the investigators hope to capture during a forced-cough recording and while sleeping can be used as biomarkers for early detection of exacerbation. These changes could be used to predict an asthma exacerbation, and provide the wearer with instant feedback allowing the user to intervene early and prevent progression to more severe symptoms. Young adults are likely to adopt wearable technologies to facilitate chronic disease management, making this an ideal age group to examine the utility of wearable devices to detect early physiologic predictors of an impending exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (14-18 years old) with asthma will be included.
* Participants will have to be diagnosed with persistent asthma (as characterized in their UNC health record) that is poorly controlled since this is the focus of the study. They will be identified as eligible for inclusion by the UNC Coordinator partner. However, they should not have any other lung disease other than asthma. They should not be taking any oral steroids every day to control their asthma. They should not need to use their asthma rescue medication multiple times a day to help with their asthma symptoms. They should not have experienced wheezing brought on when performing a lung function test.
* Participants should have Wireless Internet access at their homes
* Individuals with COVID-19 symptoms will be automatically excluded due to their clinical screening prior to their clinic visit. However, if a participant contracts COVID-19 during the study, they will be encouraged to continue participating since all interactions will be remote after the first clinical screening.
* Adolescents should be able to use a iOS device (provided by the researchers) and the devices (with assistance from parents when appropriate) for data collection efforts. They cannot participate in this study if they don't feel comfortable with operating the multiple devices including the iOS device. The iOS device can only be used for the purposes of this study. The iOS device will be restricted by enabling Parental Control Settings accessible only to the researchers.
* The participation of an adolescent may be terminated by the investigator if they do not follow the guidelines for the study, including using the devices as instructed or participating in the interviews and weekly surveys. Also, the monthly renewal for the participation of the study (up to 4 months) will be decided by the investigators on a month-by-month basis given that the participant also agrees to continue in the study.
* Individuals with physical challenges are allowed to be incidentally included as long as they satisfy all the previous criteria.

Exclusion Criteria:

* none listed

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with asthma will be included
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Identify the correlation between continuous physiological measurements, inhaler usage and lung function outcomes from spirometry | Continuously from baseline and up to 4 months
  Physiological measurements obtained from wearable devices (including motion, heart rate and heart rate variability) and from acoustic sensors (including audio from cough) will be correlated with outcomes from the daily spirometry measurements and inhaler use. Hand-crafted and data-driven features will be extracted for physiological measurements. Standard statistical tests will be used to determine significant correlations.

SECONDARY OUTCOMES:
Develop a predictive model for asthma exacerbation and drop in lung function based on physiological measurements and inhaler usage | Continuously from baseline and up to 4 months
  Results from the primary outcome will be used to build a data-driven predictive model for the detection of asthma exacerbation (as reported by the participants in their weekly survey) and drop in lung function (as measured by the spirometer). Standard metrics capturing specificity and sensitivity of the model will be used for evaluation. These models will be continuously developed after the completion of data collection from the first cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Children's Raleigh Clinic, Raleigh, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04845932/ICF_000.pdf